CLINICAL TRIAL: NCT05309798
Title: The Effect of Acute Time-Restricted Eating on Energy Intake, Subjective Appetite and Glycaemic Control in Young Healthy Males
Brief Title: Acute Time-Restricted Eating in Young Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Principal Investigator, William Mode, Principle Investigator, Nottingham Trent University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: WM_eFAST_2020
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Obesity Prevention
Keywords: Chrononutrition; Time-Restricted Eating; Energy Balance; Glycaemic Control
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: The study design is a randomised, controlled, crossover design in which participants undertake three conditions in a randomised order with at least one week in between trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Evening Fasting (Experimental): Participants will undertake acute evening fasting (feeding between 8am-4pm)
  Interventions: Behavioral: Evening Fasting
- Control (Experimental): Participants will undertake an acute standard western feeding pattern (feeding between 8am-8pm).
  Interventions: Behavioral: Control
- Morning Fasting (Experimental): Participants will undertake an acute morning fasting trial (feeding between 12pm-8pm).
  Interventions: Behavioral: Morning Fasting

INTERVENTIONS:
Behavioral: Evening Fasting — Participants will undertake acute evening fasting (feeding between 8am-4pm) for one day. After which they will attend the laboratory, following a 16 h fast, where baseline measures will be taken and the response to a standardised meal will take place. The participant will also have an opportunity to feed ad-libitum before they leave the laboratory.
  Arms: Evening Fasting
Behavioral: Morning Fasting — Participants will undertake an acute morning fasting trial (feeding between 12pm-8pm). After which, participants will visit the laboratory the following day, after a 16 h fast, where baseline measures will be taken and the response to a standardised meal will take place. The participant will also have an opportunity to feed ad-libitum before they leave the laboratory.
  Arms: Morning Fasting
Behavioral: Control — Participants will undertake an acute standard western feeding pattern (feeding between 8am-8pm). After which, participants will visit the laboratory the following day, after a 12 h fast, where baseline measures will be taken and the response to a standardised meal will take place. The participant will also have an opportunity to feed ad-libitum before they leave the laboratory.
  Arms: Control

SUMMARY:
This study compared the metabolic response to three different eating windows (morning fast,12pm-8pm; evening fast, 8am-4pm; control, 8am-8pm).

DETAILED DESCRIPTION:
Humans have evolved as a diurnal species, internally governed by the circadian system, which dictates our hormone regulation. 'Chrononutrition' is a sub-discipline which combines food timing with circadian physiology. The most popular method of time-restricted feeding in the UK is to skip breakfast. However, data from several meta-analysis have shown that skipping breakfast is associated with weight gain and insulin resistance, likely due to eating later into the evening/night and therefore, out of sync with our circadian rhythm. Recent research has shown that skipping dinner (evening fasting) has improved markers of cardio-metabolic health in clinical populations, although these are typically from longer-term studies. Despite these promising findings, it is not yet known whether these findings are population specific.

Therefore, the investigators are interested in examining the metabolic response pre and post-intervention to see whether these promising findings can translate into a healthy population. Furthermore, the investigators will be monitoring subjective appetite, energy intake, and expenditure to assess whether there is any short-term adaptation to a specific feeding window.

ELIGIBILITY:
Inclusion Criteria:

* recreationally active
* non-smokers
* non-dieting
* weight stable (self-reported for >6 months)
* were not consuming any medication known to affect appetite or physical activity

Exclusion Criteria:

* Smokers
* >10 hours per week physical activity
* Have dieted within the past 6 months
* Excessive alcohol consumption (>14 units/week)
* Use of medication or supplements that may affect hormone concentrations.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Glycaemic Control | 0 hour (Pre breakfast), 1 hour, 2 hour, 3.5 hour
  A metabolic assessment lasting 3.5 hours will take place following a standardised, laboratory-based meal. The investigators will be taking periodic capillary and venous blood samples to measure post-prandial glucose and insulin, which together comprise 'glycaemic control'.

SECONDARY OUTCOMES:
Energy Intake | 3.5 hour following breakfast
  Energy intake will be measured both during lab and outside of the laboratory when the participants are free-living. During lab, energy intake will be measured through ad-libitum feeding buffet where 20 minutes will be permitted to eat as much or as little as they desire, until 'comfortably full and satisfied', followed by post-feeding measurement of the remaining food.
Energy expenditure | Activity recorded across day 1 standardisation and day 2 (lab visit and post lab visit)
  Energy expenditure will be measured via a chest-worn device (Actiheart) which combines heart rate and accelerometry to gauge calories expended.
Visual analogue scale for subjective ratings of appetite | 0 hour (pre-breakfast), 1 hour, 2 hour, 3 hour, 4 hour (post breakfast during lab visit)
  Subjective appetite will be measured on mobile devices via a software which replicates a 100mm visual analogue scale. The scale is divided into subscales of different appetite perceptions including: hunger, fullness, desire to eat and prospective food consumption. This will be measured on a scale of 0-100 (0 - none at all) (100 - a lot).
Acylated Ghrelin (Appetite hormone) | 0 hour (pre breakfast), 1 hour, 2 hour, and 3 hour post breakfast
  Acylated Ghrelin will be measured from the venous samples taken during the post-prandial period following the standardised meal.
PYY (Appetite hormone) | 0 hour (pre-breakfast), 1 hour, 2 hour, and 3 hour post breakfast
  Acylated Ghrelin will be measured from the venous samples taken during the post-prandial period following the standardised meal.
Carbohydrate Oxidation | 0 hour (pre breakfast), 1 hour, 2 hour, 3 hour post breakfast
  Investigators will be collecting expired air into Douglas bags, and measuring the VO2 and VCO2 concentration to calculate carbohydrate oxidation.
Fat Oxidation | 0 hour (pre breakfast), 1 hour, 2 hour, 3 hour
  Investigators will be collecting expired air into Douglas bags, and measuring the VO2 and VCO2 concentration to calculate fat oxidation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Trent University, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Result] Jamshed H, Beyl RA, Della Manna DL, Yang ES, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves 24-Hour Glucose Levels and Affects Markers of the Circadian Clock, Aging, and Autophagy in Humans. Nutrients. 2019 May 30;11(6):1234. doi: 10.3390/nu11061234. PMID 31151228
- [Result] Ravussin E, Beyl RA, Poggiogalle E, Hsia DS, Peterson CM. Early Time-Restricted Feeding Reduces Appetite and Increases Fat Oxidation But Does Not Affect Energy Expenditure in Humans. Obesity (Silver Spring). 2019 Aug;27(8):1244-1254. doi: 10.1002/oby.22518. PMID 31339000
- [Result] Hutchison AT, Regmi P, Manoogian ENC, Fleischer JG, Wittert GA, Panda S, Heilbronn LK. Time-Restricted Feeding Improves Glucose Tolerance in Men at Risk for Type 2 Diabetes: A Randomized Crossover Trial. Obesity (Silver Spring). 2019 May;27(5):724-732. doi: 10.1002/oby.22449. Epub 2019 Apr 19. PMID 31002478
- [Result] Templeman I, Gonzalez JT, Thompson D, Betts JA. The role of intermittent fasting and meal timing in weight management and metabolic health. Proc Nutr Soc. 2020 Feb;79(1):76-87. doi: 10.1017/S0029665119000636. Epub 2019 Apr 26. PMID 31023390
- [Result] Popkin BM. The nutrition transition and obesity in the developing world. J Nutr. 2001 Mar;131(3):871S-873S. doi: 10.1093/jn/131.3.871S. PMID 11238777
- [Result] Allison KC, Goel N. Timing of eating in adults across the weight spectrum: Metabolic factors and potential circadian mechanisms. Physiol Behav. 2018 Aug 1;192:158-166. doi: 10.1016/j.physbeh.2018.02.047. Epub 2018 Feb 24. PMID 29486170
- [Result] St-Onge MP, Ard J, Baskin ML, Chiuve SE, Johnson HM, Kris-Etherton P, Varady K; American Heart Association Obesity Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular Disease in the Young; Council on Clinical Cardiology; and Stroke Council. Meal Timing and Frequency: Implications for Cardiovascular Disease Prevention: A Scientific Statement From the American Heart Association. Circulation. 2017 Feb 28;135(9):e96-e121. doi: 10.1161/CIR.0000000000000476. Epub 2017 Jan 30. PMID 28137935